CLINICAL TRIAL: NCT00809367
Title: Collection and Banking of Leukemia Cells for Vaccine Generation and Research in Patients With Advanced MDS or AML
Brief Title: Collection and Banking of Leukemia Cells MDS/AML
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Vincent T. Ho, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 08-159
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-01

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloid Leukemia
Keywords: MDS; AML; banking study
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Collection of Leukemia Cells (Other): Other: Collection of Leukemia Cells Collection of leukemia cells either by 1) routine blood draw 2) bone marrow aspirate or 3) leukopheresis
  Interventions: Other: Collection of Leukemia Cells

INTERVENTIONS:
Other: Collection of Leukemia Cells — Collection of leukemia cells either by 1) routine blood draw 2) bone marrow aspirate or 3) leukopheresis

SUMMARY:
The goal of this research study is to determine if it is feasible to collect leukemia cells from patients ahead of time (before they undergo further treatments) so that these cells (after being radiated so they will no longer grow or divide) can be given back to them as a cancer vaccine if/after the participant receives a bone marrow or blood stem cell transplant in the future. The purpose of the research study will be to collect, freeze and store leukemia calls from participants blood or bone marrow. This study is a companion study to a vaccine study.

DETAILED DESCRIPTION:
* Leukemia cells will be collected by one or more of the following methods: 1)Routine blood draw 2)Bone marrow aspirate 3) Leukapheresis. The physician and study staff will determine which of the methods above is best suited for each participant.
* After collection, the leukemia cells will be transported to the Cell Manipulation Core Facility (CMCF) at the Dana-Farber Cancer Institute, where they will be frozen until the time of vaccine administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML will be eligible for banking at the time of relapse or primary induction failure or at the time of AML diagnosis they are 60 years of age or older, AML arising out of background MDS or MPD or AML known with high risk cytogenetics
* Patients with MDS-RAEB-1 or RAEB-II, CMML-1 or CMML-II
* Patients must have >5% blast in bone marrow or peripheral blood
* ECOG Performance Status 0-2
* Age greater than or equal to 18 years
* Reasonable likelihood, in the physician's opinion, that the patient will be a candidate for allogeneic stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of banking leukemic blood or marrow samples from patients with advanced MDS or AML such that these cells could be used for tumor cell vaccination at a later date. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Ho, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States